CLINICAL TRIAL: NCT05544058
Title: Retrospective Non-interventional Study of Stiripentol Use in Dravet Patients in the USA
Status: Completed | Type: Observational
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Other Study IDs: STIRUS (STP228)
Record Dates: First submitted 2022-08-24; First posted 2022-09-16 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Dravet Syndrome
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective study — Retrospective study

SUMMARY:
The present study aims to collect data regarding the history of the disease, previous and current treatments, and the clinical status of Dravet patients during the 3 months prior to stiripentol initiation, the first 3 months on stiripentol and the last 3 months on stiripentol (irrespective of stiripentol discontinuation).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Dravet syndrome
* Treated with stiripentol for a minimum of 3 months in routine practice

Exclusion Criteria:

* NA

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patient with dravet syndrome and reated with stiripentol for a minimum of 3 months in routine practice
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
management of the Dravet syndrome | through study completion, an average of 1 year
  Patient Information History of the Disease Clinical status of the patient during the 3 months preceding stiripentol treatment initiation Clinical status of the patient at stiripentol initiation Clinical status of the patient during the first 3 months of stiripentol treatment Clinical status of the patient during the last 3 months of stiripentol treatment Evolution on stiripentol

SECONDARY OUTCOMES:
Better detection of the Dravet syndrome | through study completion, an average of 1 year
  Patient Information History of the Disease Clinical status of the patient during the 3 months preceding stiripentol treatment initiation Clinical status of the patient at stiripentol initiation Clinical status of the patient during the first 3 months of stiripentol treatment Clinical status of the patient during the last 3 months of stiripentol treatment Evolution on stiripentol

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No